CLINICAL TRIAL: NCT00005972
Title: Phase II Trial of Gemcitabine/Irinotecan as Second Line Therapy for Small Cell Lung Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Recurrent or Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-39902; U10CA031946 (NIH); CALGB-39902; CDR0000067959 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-07-05; First posted 2004-03-24 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine + irinotecan (Experimental): Patients are stratified according to prior response duration (progression 90 days or more after initial therapy vs progression less than 90 days after initial therapy or no response to initial therapy). Patients receive gemcitabine IV over 30 minutes and irinotecan IV over 90 minutes on days 1 and 8. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 1 year, then every 6 months for 2 years, and then annually for 3 years.
  Interventions: Drug: gemcitabine hydrochloride; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have recurrent or refractory small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the overall, complete, and partial response rates of patients with recurrent or refractory small cell lung cancer when treated with gemcitabine plus irinotecan. II. Determine the overall and failure free survival of these patients when treated with this regimen. III. Determine the duration of response of these patients after this treatment. IV. Evaluate the toxicity associated with the administration of this treatment in this patient population.

OUTLINE: Patients are stratified according to prior response duration (progression 90 days or more after initial therapy vs progression less than 90 days after initial therapy or no response to initial therapy). Patients receive gemcitabine IV over 30 minutes and irinotecan IV over 90 minutes on days 1 and 8. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 1 year, then every 6 months for 2 years, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 78 patients will be accrued for this study over 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed recurrent or refractory small cell lung cancer Measurable disease At least 20 mm with conventional techniques OR At least 10 mm with spiral CT scan The following are not considered measurable: Bone lesions Leptomeningeal disease Ascites Pleural/pericardial effusion Abdominal masses not confirmed and followed by imaging techniques Cystic lesions Tumor lesions situated in a previously irradiated area Known CNS metastases allowed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: CTC 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception No prior or concurrent malignancy in past 5 years except curatively treated carcinoma in situ of the cervix, breast, or basal cell or squamous cell carcinoma of the skin

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No more than 1 prior chemotherapy or chemoradiotherapy regimen No prior gemcitabine or irinotecan Endocrine therapy: Not specified Radiotherapy: No more than 1 prior chemoradiotherapy regimen At least 2 weeks since prior cranial radiotherapy for CNS metastases No concurrent cranial radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2000-05; Primary Completion 2006-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
overall response rate | Up to 18 weeks

SECONDARY OUTCOMES:
overall survival | Up to 18 weeks
failure-free survival | Up to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Caio Max Rocha Lima, MD, Study Chair — Medical University of South Carolina
Locations (50):
- United States (50):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Rocha-Lima CM, Herndon JE 2nd, Lee ME, Atkins JN, Mauer A, Vokes E, Green MR; Cancer and Leukemia Group B. Phase II trial of irinotecan/gemcitabine as second-line therapy for relapsed and refractory small-cell lung cancer: Cancer and Leukemia Group B Study 39902. Ann Oncol. 2007 Feb;18(2):331-7. doi: 10.1093/annonc/mdl375. Epub 2006 Oct 25. PMID 17065590